CLINICAL TRIAL: NCT06774326
Title: Role of Spectral CT in the Evaluation of Cardiotoxicity in Patients With Hodgkin's Lymphoma and Diffuse Large B-cell Lymphoma Treated With Anthracyclines
Acronym: AntraCardioTox
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: AntraCardioTox Linfoma Spectra
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Imaging; Cardiac Imaging Techniques; Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Lymphoma; Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the diagnostic capability of Spectral CT (performed with contrast agent as part of routine oncological follow-up) in detecting signs of acute and chronic early-onset cardiac toxicity from anthracyclines in patients with Hodgkin's lymphoma and diffuse large B-cell lymphoma undergoing treatment regimens that include a drug from this family.

DETAILED DESCRIPTION:
To evaluate the diagnostic capability of Spectral CT, performed with contrast agent during routine oncological follow-ups, in detecting signs of acute and chronic early-onset cardiac toxicity caused by anthracyclines in patients with Hodgkin's lymphoma and diffuse large B-cell lymphoma undergoing treatment regimens including anthracycline-based drugs. Spectral CT provides advanced data, such as iodine maps and tissue characterization, allowing for the identification and quantification of hyperemia, edema, and fibrosis. These findings are particularly promising in cardiovascular imaging, where tissue characterization and early detection of myocardial damage (edema or fibrosis) are traditionally achieved with cardiac MRI (cardio-MRI).

In clinical oncology, anthracyclines improve survival rates but are associated with cardiotoxic effects, classified as acute (up to two weeks after therapy), early chronic (within one year), or late chronic (years or decades later), often irreversible. Anthracycline-related cardiac toxicity is dose-dependent and varies from subclinical alterations to overt symptoms such as arrhythmias, fibrosis, and heart failure. Early detection of myocardial damage with imaging techniques is critical for initiating cardioprotective therapy, which can significantly improve cardiac outcomes.

Currently, functional imaging modalities like echocardiography and cardio-MRI are used. While echocardiography offers functional data such as LVEF and strain, cardio-MRI provides more precise and reproducible measurements and structural data (e.g., edema via T2 mapping and fibrosis via late gadolinium enhancement, LGE). Structural markers, such as positive LGE and elevated T1 mapping or ECV values, are highly sensitive and can detect damage before functional decline, enabling earlier intervention. However, cardio-MRI has limitations, such as long acquisition times, high costs, and contraindications like claustrophobia.

With the introduction of Spectral CT, studies have shown that advanced CT scanners can also visualize and quantify myocardial fibrosis (as late-iodine enhancement, LIE) and measure ECV, comparable to cardio-MRI. This suggests that Spectral CT could become a "one-stop-shop" modality, capable of assessing both the patient's primary disease and signs of anthracycline-induced cardiotoxicity through post-processing of the same images, even in subclinical stages.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Hodgkin's lymphoma or diffuse large B-cell lymphoma (DLBCL) undergoing treatment regimens including anthracyclines
* Age ≥18 years
* Informed consent obtained

Exclusion Criteria:

* Absolute or relative contraindications to CT examination and/or administration of iodinated contrast agents (e.g., pregnancy, severe renal insufficiency in non-dialysis patients with GFR <15-30 ml/min/1.73m²).
* Patients with a concomitant positive history of cardiovascular disease (e.g., myocardial infarction, known coronary artery disease, heart failure, arrhythmias, prior myocarditis, cardiomyopathies).
* History of mediastinal radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Hodgkin's lymphoma and diffuse large B-cell lymphoma (DLBCL) undergoing treatment regimens including anthracyclines will participate in the study. They will be enrolled and undergo CT and MRI follow-ups conducted by the cardiac radiology team.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Myocardial damage | 36 months after starting CHT
  Diagnosis of the presence of acute myocardial damage (hyperemia present) or chronic damage (hyperemia absent) based on the evaluation of the following parameters obtained from Spectral CT:
  * Increased ECV (ECV value above the upper limit of normality, set at 30%).
  * Presence of Late Iodine Enhancement (LIE) in the myocardium (areas of myocardial hyperdensity due to late-phase iodine contrast accumulation) and its relative extent.
  * Presence of Hyperemia or Hypoperfusion using the Spectral "Iodine No Water" parameter (visual scoring of hyper- or hypodense areas; consideration of a possible quantitative score in mgI/ml).
  * Diagnosis of myocardial damage due to chemotherapy (CHT) based on clinical practice upon hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russo, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No